CLINICAL TRIAL: NCT06292962
Title: Evaluating the Impact of Vagus Nerve Stimulation on Diabetic Peripheral Neuropathic Pain - A Randomized, Double-Blinded, Sham-Controlled Study
Brief Title: Evaluating the Impact of Vagus Nerve Stimulation on Diabetic Peripheral Neuropathic Pain
Acronym: VNSDPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saima Abass Tahammal (Other)
Collaborators: Al Ain University (Unknown)
Responsible Party: Sponsor-Investigator, Saima Abass Tahammal, Principal Investigator, Shifa International Hospital
Organization: Shifa International Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SH-34988389
Record Dates: First submitted 2023-12-24; First posted 2024-03-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathies; Type2diabetes; Neuropathic Pain
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a randomized, double-blinded, sham-controlled, parallel group clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group VTG (Experimental): Group VTG will receive active non-invasive transcutaneous vagal nerve stimulation (tVNS)
  Interventions: Device: non-invasive transcutaneous vagal nerve stimulation (tVNS)
- Group STG (Sham Comparator): Group STG will receive Inactive sham stimulation
  Interventions: Device: Sham device

INTERVENTIONS:
Device: non-invasive transcutaneous vagal nerve stimulation (tVNS) — The device is used stimulate the vagus nerve
  Other Names: tVNS device
  Arms: Group VTG
Device: Sham device — Sham device that does not stimulate the vagus nerve
  Other Names: SD
  Arms: Group STG

SUMMARY:
The purpose of the study is to investigate the effects of non-invasive invasive vagal nerve stimulation on diabetic peripheral neuropathic pain in people with diabetes.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded, sham-controlled, parallel-group clinical trial, which will include participants with diabetic peripheral neuropathic pain.

Participants are randomized to receive either active non-invasive transcutaneous vagal nerve stimulation (tVNS) or inactive sham stimulation.

The study will investigate the effects of short-term, high-intensity tVNS treatment on peripheral pain.

The primary outcome is subjective patient evaluation of pain symptoms by the use of validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes mellitus > 1 year
* Patients experiencing neuropathic pain

Exclusion Criteria:

* Patients with co-morbidities such as chronic pain from other conditions
* Patients with serious complications of diabetes such as nephropathy and retinopathy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Neuropathic pain scores | up to 24 weeks
  Change in neuropathic pain scores assessed by validated questionnaire

SECONDARY OUTCOMES:
Quality of life score | up to 24 weeks
  Patient's perception of quality of life assessed by validated questionannaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shifa Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No